CLINICAL TRIAL: NCT00738439
Title: Prospective, Multi-Center Adult Spinal Deformity Outcomes Database Registry
Acronym: PON
Status: Active, not recruiting | Type: Observational
Sponsor: Shay Bess (Other)
Collaborators: DePuy Spine (Industry); K2M, Inc. (Industry); NuVasive (Industry); Zimmer Biomet (Industry); Orthofix Inc. (Industry)
Responsible Party: Sponsor-Investigator, Shay Bess, President, ISSGF, International Spine Study Group Foundation
Organization: International Spine Study Group Foundation (Other)
Other Study IDs: 1-08-1850
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Spinal Deformity
Keywords: scoliosis; kyphosis; treatment outcomes; spinal deformity
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Operative: Diagnosis of adult degenerative or idiopathic scoliosis with a curvature of the spine measuring greater than or equal to 20 degrees requiring surgery.
- Nonoperative: Diagnosis of adult degenerative or idiopathic scoliosis with a curvature of the spine measuring greater than or equal to 20 degrees not requiring surgery.

SUMMARY:
The clinical, radiographic, and HRQL outcomes will be compared in operative and nonoperative adult spinal deformity patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult degenerative or idiopathic scoliosis with a curvature of the spine measuring greater than or equal to 20 degrees
* Sagittal Vertical Axis (SVA) > 5cm
* Pelvic Tilt > 25 degrees
* Thoracic kyphosis > 60 degrees
* Age 18 or greater at the time of enrollment.

Exclusion Criteria:

* Diagnosis of scoliosis other than degenerative or idiopathic (i.e. paralytic/neuromuscular, congenital)
* Age <18 yrs at time of surgery or initial consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater than 18 years of age who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1999 (Actual)
Dates: Start 2008-10; Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic | initial visit, 1 year, 2 years, 3-5 years
  Coronal and Sagittal views of the spine

SECONDARY OUTCOMES:
Clinical outcomes | initial visit, 1 year, 2 years, 3-5 years
  physical examination/pain scale
Health related quality of life | initial visit, 1 year, 2 years, 3-5 years
  Oswestry, SRS22r, SF-36, LSDI, EQ5D3L, NDI DRAM (optional)

CONTACTS AND LOCATIONS:
Overall Officials: Shay Bess, MD, Principal Investigator — Denver International Spine Center
Locations (9):
- United States (9):
  - Scripps Clinic, La Jolla, California
  - University of California - Davis, Sacramento, California
  - University of California - San Francisco Medical Center, San Francisco, California
  - Denver International Spine Center, Denver, Colorado
  - Doug Burton, MD, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - NYU Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Passias PG, Soroceanu A, Scheer J, Yang S, Boniello A, Smith JS, Protopsaltis T, Kim HJ, Schwab F, Gupta M, Klineberg E, Mundis G, Lafage R, Hart R, Shaffrey C, Lafage V, Ames C; International Spine Study Group. Magnitude of preoperative cervical lordotic compensation and C2-T3 angle are correlated to increased risk of postoperative sagittal spinal pelvic malalignment in adult thoracolumbar deformity patients at 2-year follow-up. Spine J. 2015 Aug 1;15(8):1756-63. doi: 10.1016/j.spinee.2015.04.007. Epub 2015 Apr 8. PMID 25862507